CLINICAL TRIAL: NCT04519996
Title: Pre-operative Ultrasonographic Evaluation of the Internal Jugular Vein Collapsibility Index and Inferior Vena Cava Collapsibility Index to Predict Post Spinal Hypotension in Pregnant Women Undergoing Caesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amr Arafa Elbadry, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IJVCI versus IVCCI
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-08

CONDITIONS: Cesarean Section
Keywords: cesarean section; hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US Internal Jugular Vein Collapsibility Index (Experimental): The US transducer will be placed on the right side of the neck in the transverse plane over RIJV 2 cm above the sternoclavicular joint. The IJV will be identified by the color flow Doppler and compressibility.
  Interventions: Procedure: US Internal Jugular Vein Collapsibility Index measurment
- US Inferior Vena Cava Collapsibility Index (Experimental): The transducer will be placed in the subxiphoid region in a longitudinal position. IVC measurements will be made just distal to the IVC-hepatic vein junction, approximately 3 to 4 cm distal to the right atrium. The IVC will be identiﬁed by Doppler waveform, compressibility and phasic collapse with respiration.
  Interventions: Procedure: US Inferior Vena Cava Collapsibility Index measurment

INTERVENTIONS:
Procedure: US Internal Jugular Vein Collapsibility Index measurment — Machine
  A sonosite M-Turbo ultrasound machine will be used for all the examinations. A curvilinear USG probe for IVC imaging (1-5 MHz, 21 mm).
  The US transducer will be placed on the right side of the neck in the transverse plane over RIJV 2 cm above the sternoclavicular joint. The IJV will be identified by the color flow Doppler and compressibility. Care will be taken not to compress or obliterate the vein by applying minimal pressure. When the whole circumference of the vein will be visible the measurements were done. The recordings will be done for four respiratory cycles. The maximum, minimum AP diameters, and cross-sectional area will be estimated and, from this, corresponding CI will be derived (Maximum diameter or cross-sectional area (CSA)-minimum diameter or CSA/maximum diameter or CSA) ×100%. All the above measurements will be repeated with the head end of patients elevated to 30° position.
  Arms: US Internal Jugular Vein Collapsibility Index
Procedure: US Inferior Vena Cava Collapsibility Index measurment — Machine
  A sonosite M-Turbo ultrasound machine will be used for all the examinations. A linear vascular transuder for IJV imaging (7-13 MHz, 38 mm) will be used.
  The transducer will be placed in the subxiphoid region in a longitudinal position. IVC measurements will be made just distal to the IVC-hepatic vein junction, approximately 3 to 4 cm distal to the right atrium. The IVC will be identiﬁed by Doppler waveform, compressibility and phasic collapse with respiration. The maximum (IVCD) and minimum (IVCD) internal anteroposterior (AP) diameters of the IVC at the end of expiration and inspiration respectively over the same respiratory cycle will be measured. The IVCCI is derived from the equation, IVCCI= (IVCD max -IVCD min)/IVCD max × 100.
  Arms: US Inferior Vena Cava Collapsibility Index

SUMMARY:
Postspinal hypotension (PSH) is common in obstetric anesthesia practice, with an incidence of up to 71 %. PSH can occur precipitously and, if severe, can result in both maternal and fetal/neonatal adverse events. Pregnant women with predelivery hypovolemia are at risk of cardiovascular collapse and the sympathetic blockade may severely decrease venous return. Hence, prevention of PSH is an essential element in obstetric anesthesia and fasting for aspiration prophylaxis may further add up to the hypovolemia for the patients not on maintenance fluids.

Hemodynamic monitoring in obstetric patients has evolved during the last decade, with the development of minimally invasive and noninvasive continuous cardiac output (CO) monitors. Ultrasound (USG) is a method for noninvasive hemodynamic optimization in the ICU and ED, and it may be more helpful than other noninvasive methods. Transabdominal USG measurements of inferior vena cava (IVC) are noninvasive and thus are not associated with complications. USG of the IVC diameter is a useful and easy method for assessing a patient's volume status by calculating the IVC collapsibility index (IVCCI).

Recently, the usefulness of point-of-care ultrasonographic examination, performed by anesthesiologists in real time, for perioperative management has been reported . Ultrasonographic studies have established the utility of measuring the inferior vena cava (IVC) or internal jugular Vein (IJV) for evaluating intravascular volume status .

In particular, IVC diameter and collapsibility, obtained from ultrasonographic measurement, have been demonstrated to be predictors of hypotension after anesthetic administration.

DETAILED DESCRIPTION:
Pregnant women planned for elective surgery will be advised for nil per oral after midnight and. After detailed preanesthetic checkup, on arrival in operating room, standard monitoring devices will be attached (pulse oximeter, noninvasive blood pressure and 3-lead electrocardiography).

Machine

A sonosite M-Turbo ultrasound machine will be used for all the examinations. A curvilinear USG probe for IVC imaging (1-5 MHz, 21 mm). A linear vascular transuder for IJV imaging (7-13 MHz, 38 mm) will be used.

Measurements

IJV measurement

All the measurements will be done on Right IJV with the patients initially lying supine at 0° and later head end elevated at 30°. With the patients in supine position, the USG transducer will be placed on the right side of the neck in the transverse plane over RIJV 2 cm above the sternoclavicular joint. The IJV will be identified by the color flow Doppler and compressibility. Care will be taken not to compress or obliterate the vein by applying minimal pressure. When the whole circumference of the vein will be visible the measurements were done. The recordings will be done for four respiratory cycles. The maximum, minimum AP diameters, and cross-sectional area will be estimated and, from this, corresponding CI will be derived (Maximum diameter or cross-sectional area (CSA)-minimum diameter or CSA/maximum diameter or CSA) ×100%. All the above measurements will be repeated with the head end of patients elevated to 30° position

IVC measurements

The transducer will be placed in the subxiphoid region in a longitudinal position. IVC measurements will be made just distal to the IVC-hepatic vein junction, approximately 3 to 4 cm distal to the right atrium. The IVC will be identiﬁed by Doppler waveform, compressibility and phasic collapse with respiration. The maximum (IVCD) and minimum (IVCD) internal anteroposterior (AP) diameters of the IVC at the end of expiration and inspiration respectively over the same respiratory cycle will be measured. The IVCCI is derived from the equation, IVCCI= (IVCD max -IVCD min)/IVCD max × 100.

The patients will be positioned in sitting position to give the spinal anesthesia at L3-L4/L2-L3 intervertebral level in the midline approach. After local infiltration of skin and subcutaneous tissue with 2% lignocaine, 25 G B-braun spinal needle will be used to administer subarachnoid block (SAB) with 2.5 ml of hyperbaric bupivacaine (5%) and 20 µg of fentanyl after confirmation of free flow of cerebrospinal fluid (CSF) at the hub of the needle. Patients will be coloaded with 10-12 ml/kg (over the period of 15 min) of Ringer's Lactate (RL) solution at the time of SAB. Thereafter, patients will be placed in supine position with wedge under the right hip. HR, systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), and SpO2 will be recorded throughout the procedure every 3 min till 15 min of SAB. Level of sensory block will be assessed by response to cold touch and surgery will be allowed after sensory blocks reaches to T6 level. Hypotension (reduction in MAP more than 20% and/or MAP <65 mmHg) will be treated with 6 mg of injection of ephedrine and a bolus of 250 ml of Ringer's Lactate (RL) solution over 10 minutes. Number of boluses of ephedrine and fluids will be recorded. Bradycardia (Heart Rate < 50 beats/ min) will be treated with 0.6 mg of injection atropine.

Data collection

The attending anaesthesiologist who will perform subarachnoid block (SAB) and will monitor the patient during the study period will be blinded to the ultrasound measurements of both inferior vena cava collapsibility index (IVCCI) and internal jugular vein collapsibility index (IJVCI) which will be recorded by either of the two investigators pre-operatively.

Measurements:

1. Demographic data as age, weight, height and ASA status.
2. Hemodynamics including heart rate, mean arterial blood pressure every 3 min till 15 min of SAB.
3. Number of boluses of ephedrine and fluids will be recorded
4. Inferior vena cava collapsibility index (IVCCI) and internal jugular vein collapsibility index (IJVCI).

ELIGIBILITY:
Inclusion Criteria:

1.55 female patients 2. aged 20-40 years 3.ASA Physical Status Class I and II 4. scheduled for elective lower segment cesarean section

Exclusion Criteria:

1. Patients who will refuse
2. Emergency LSCS
3. Patients with expected massive intraoperative blood loss e.g. placenta Previa and placenta accreta
4. Cardiovascular, respiratory, renal diseases
5. Patients who will receive preloading of intravenous fluid

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 55 (Estimated)
Dates: Start 2020-10-30 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
pre-operative inferior vena cava collapsibility index (IVCCI) | pre-operative
  for predicting post-spinal anaesthesia hypotension (PSAH). The maximum (IVCD) and minimum (IVCD) internal anteroposterior (AP) diameters of the IVC at the end of expiration and inspiration respectively over the same respiratory cycle will be measured. The IVCCI is derived from the equation, IVCCI= (IVCD max -IVCD min)/IVCD max × 100
pre-operative internal jugular vein collapsibility index (IJVCI) | pre-operative
  for predicting post-spinal anaesthesia hypotension (PSAH), The maximum, minimum antero-pestorior diameters, and cross-sectional area will be estimated and, from this, corresponding collapsibility index will be derived (Maximum diameter or cross-sectional area (CSA)-minimum diameter or CSA/maximum diameter or CSA) ×100%.

IPD SHARING:
Plan to Share IPD: No